CLINICAL TRIAL: NCT00826189
Title: A Follow-up Study to 7 Years of a Randomized, Double-blinded, Placebo-controlled Study on the Influence of Probiotics on Atopy With Focus on Respiratory Allergic Diseases
Brief Title: Influence of Probiotics on Atopy With Focus on Respiratory Allergic Diseases- Follow-up to 7 Years
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Paediatrics, A/Prof Lynette Shek, National University Hospital, Singapore
Other Study IDs: SQNU01 (Phase III)
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: Probiotics; Asthma; Allergic Rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators had conducted an initial double-blind, placebo-controlled clinical trial (NCT00318695) to study the effects of probiotic supplementation from birth to 6 months of age in the incidence of atopic diseases at 2 years old. This is then further investigated up to 5 years of age in a follow-up study NCT00365469 to assess the longer term beneficial effects.

This current study intends to follow-up for another 2 years until 7 years of age as this is critical in the evaluation of respiratory allergies in the form of clinical asthma and allergic rhinitis.

DETAILED DESCRIPTION:
This study intends to continue the initial double-blind, placebo-controlled randomized clinical trial (NCT00318695) which involved 253 subjects with a first degree family history of allergic disease. The infants received at least 60ml of commercially available cow's milk based infant formula with or without probiotic supplementation (Bifidobacterium longum [BL999] 1×10*7 colony-forming unit (cfu)/g and Lactobacillus rhamnosus [LPR]2×10*7 cfu/g) daily from the first day of life for the first 6 months. A follow-up study (NCT00365469) up to 5 years of age is currently in process.

This current study plans to continue the follow-up for a further 2 years till the cohort reaches 7 years of age. This study will only involve telephone calls which will be conducted every 3 months to ascertain for symptoms and incidence of respiratory allergic disease.This is critical in the evaluation of asthma and allergic rhinitis which tend to develop later in life and this step-wise, temporal development of respiratory allergies has been described as "Atopic March".

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the both NCT00318695 and NCT00365469 studies.
* Parent(s) / Guardian consent to the subject's participation in the study.
* Subject and the parent(s)/ guardian are willing to comply with the study procedures

Exclusion Criteria:

* The parent is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained.
* The parent is unable/ unwilling to comply with study procedures

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The subjects who have completed NCT00318695 and NCT00365469 studies will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Asthma | 7 years of age

SECONDARY OUTCOMES:
Allergic Rhinitis | 7 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Lynette Shek, A/Prof, Principal Investigator — National University Hospital, Singapore; Marion Aw, A/Prof, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore